CLINICAL TRIAL: NCT00567658
Title: Effect of Aggressive Acid Suppression With Esomeprazole on Vocal Cord Granulomas: Randomized Placebo-Controlled Trial
Brief Title: Effect of Acid Suppression With Esomeprazole on Vocal Cord Granulomas
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision of terminate the study was reached due to difficulties surrounding recruitment and enrollment of subjects since the inception of the study.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 070730
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Larynx Disease
MeSH Terms: conditions — Laryngeal Diseases | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A 1 (Placebo Comparator): Arm I: placebo group receives BID placebo
  Interventions: Drug: Esomeprazole
- A2 (Experimental): subjects receive active drug, esomeprazole 40 mg BID
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole or Nexium 40 mg BID is given for four months.

SUMMARY:
The purpose of this research study is to measure the effects of the drug, esomeprazole 40 mg (Nexium) or placebo (inactive drug) on vocal cord granulomas.

DETAILED DESCRIPTION:
Vocal cord granulomas (VCG) are common structural lesions of vocal cords attributed to vocal abuse / misuse and recently to gastroesophageal reflux. Vocal process granulomas are reactive/reparative process, in which an intact or ulcerated squamous epithelium is underlaid by granulation tissue or fibrosis (4, 5). Ulualp et al (6) have reported a higher prevalence of pharyngeal acid reflux (PAR) events in patients with vocal cord lesions. In a case control study they showed that the prevalence of pharyngeal reflux, documented with 3 site pharyngoesophageal pH monitoring, is higher among patients with posterior laryngitis and vocal cord lesions than control (78% vs. 21%). Most recently our cohort trial in over 80 patients with laryngeal findings suggestive of GERD suggested that vocal cord abnormalities such as granulomas may be more specific sign of GERD than any other (7). Thus, there is reasonable scientific intrigue regarding this laryngeal finding and the causal role from gastroesophagopharyngeal acid reflux requiring better studies. However, no study has evaluated the potential causal association between GERD and VCGs.

ELIGIBILITY:
Inclusion Criteria:

Patients with vocal cord granulomas

Exclusion Criteria:

* Age < 18
* Pregnancy
* Use of proton pump inhibitor (PPI) within the last 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
• Primary outcome: Vocal cord granuloma improvement +/- resolution Outcome categories-subjectively assessed at laryngoscopy (current practice) | 4 months

SECONDARY OUTCOMES:
Symptom improvement +/- resolution | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD, PhD, MS epi, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States